CLINICAL TRIAL: NCT04469101
Title: Which Position is Best: A Randomized Clinical Trial on the Effect That Position Has on Walking Labour Epidural Analgesia
Brief Title: A Study on the Effect of Position on Walking Labour Epidural Efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Monica San Vicente, Principal Investigator, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Bio 1813
Record Dates: First submitted 2020-06-30; First posted 2020-07-13 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Labor Pain; Analgesia, Epidural
Keywords: Analgesia, Obstetrical; Posture; Pregnancy; Female; Heart Rate, Fetal; Hypotension
MeSH Terms: conditions — Labor Pain; Agnosia; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Left Uterine Displacement (Experimental): Supine with left tilt for uterine displacement
  Interventions: Procedure: Lumbar Epidural
- Left Lateral (Experimental): Left lateral decubitus position
  Interventions: Procedure: Lumbar Epidural
- Right Lateral (Experimental): Right lateral decubitus position
  Interventions: Procedure: Lumbar Epidural
- Upright (Experimental): Upright seated position
  Interventions: Procedure: Lumbar Epidural

INTERVENTIONS:
Procedure: Lumbar Epidural — Parturients will have an epidural placed in the upright seated position as per institution standard. After epidural placement, they will be positioned as per their randomization. They will then have a total of 20 cc of epidural solution (0.08% ropivacaine with 2 mcg per cc of fentanyl) injected into the epidural in boluses of 5 cc every 5 minutes.

SUMMARY:
This study is being done to better understand how patient positioning can affect pain relief after an epidural. In addition to pain, the investigators will assess how position affects epidural spread, and its effects on maternal blood pressure and fetal heart rate.

DETAILED DESCRIPTION:
Epidurals will be placed with parturients in the standard sitting position. An epidural catheter will be placed to a depth of 5 cm into the epidural space. After placement, parturients will be randomized to one of the four position groups (left uterine displacement, left lateral, right lateral, or seated upright). After successful positioning, a series of 5 cc bolus doses of 0.08% ropivacaine with 2 mcg per cc of fentanyl will be injected through the epidural catheter in 5 minute intervals for a total volume of 20 cc. After the initial loading dose of epidural solution has been injected in the first 20 minutes post-insertion, the patient will be able to return to whatever position they are most comfortable with. The parturient will be asked to rate their pain on a verbal pain scale of between 0 and 10 at the peak of their contraction at three time intervals. The spread of the blockade will be assessed with ice applied along both the left and right mid-clavicular lines. Maternal blood pressure will be measured on the upper arm in all patients as per nursing protocol. Fetal heart rate will be monitored intermittently with Doppler ultrasound as per nursing protocol.

ELIGIBILITY:
Inclusion Criteria:

* Active labour or admitted for induction of labour
* Requesting an epidural for labour analgesia
* Contractions occurring greater than once every 5 minutes

Exclusion Criteria:

* Coagulation disorder
* High risk pregnancy as per obstetrics
* Spinal pathology (included scoliosis, herniated disks, or previous lumbar back surgery)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Labour pain based on verbal rating pain scale | Taken at time 0 minutes after epidural insertion
  Pain with contractions, assessed using a 0 to 10 verbal rating pain scale; 0 being no pain with a contraction and 10 being the worse pain with a contraction.
Labour pain based on verbal rating pain scale | Taken at time 20 minutes after epidural insertion
  Pain with contractions, assessed using a 0 to 10 verbal rating pain scale; 0 being no pain with a contraction and 10 being the worse pain with a contraction.
Labour pain based on verbal rating pain scale | Taken at time 40 minutes after epidural insertion
  Pain with contractions, assessed using a 0 to 10 verbal rating pain scale; 0 being no pain with a contraction and 10 being the worse pain with a contraction.

SECONDARY OUTCOMES:
Assessment of epidural levels based on dermatomes | Taken at time 20 minutes after epidural insertion
  Levels of analgesia assessed via temperature insensitivity to ice on the right and left side along the midclavicular lines of the patient and reported as dermatome levels.
Assessment of epidural levels based on dermatomes | Taken at time 40 minutes after epidural insertion
  Levels of analgesia assessed via temperature insensitivity to ice on the right and left side along the midclavicular lines of the patient and reported as dermatome levels.
Category of epidural based on bilateral dermatome levels | Taken at time 20 minutes after epidural insertion
  Epidural assessed if it is successful, unilateral (more than two dermatome level difference between sides), patchy (one or more areas between dermatomes that remain sensitive to temperature assessment), or failed (no measurable dermatome levels) based on the dermatome levels gathered by nursing assessments.
Category of epidural based on bilateral dermatome levels | Taken at time 40 minutes after epidural insertion
  Epidural assessed if it is successful, unilateral (more than two dermatome level difference between sides), patchy (one or more areas between dermatomes that remain sensitive to temperature assessment), or failed (no measurable dermatome levels) based on the dermatome levels gathered by nursing
Events of maternal hypotension after epidural placement | Blood pressure taken with a non-invasive blood pressure monitoring cuff every 5 minutes for 20 minutes after epidural insertion
  Hypotensive events defined as a deviation of greater than 20% of maternal blood pressure compared to pre-epidural baseline.
Events of fetal bradycardia after epidural placement | Intermittent fetal heart rate monitoring via doppler as per nursing protocol for 20 minutes after epidural insertion
  Fetal bradycardic events defined as a fetal heart rate of less than 120 bpm after epidural placement.

CONTACTS AND LOCATIONS:
Overall Officials: Monica San Vicente, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Jim Pattison Children's Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halpern SH, Walsh V. Epidural ropivacaine versus bupivacaine for labor: a meta-analysis. Anesth Analg. 2003 May;96(5):1473-1479. doi: 10.1213/01.ANE.0000052383.01056.8F. PMID 12707152
- [Background] Epidural and Position Trial Collaborative Group. Upright versus lying down position in second stage of labour in nulliparous women with low dose epidural: BUMPES randomised controlled trial. BMJ. 2017 Oct 18;359:j4471. doi: 10.1136/bmj.j4471. PMID 29046273
- [Background] Husemeyer RP, White DC. Lumbar extradural injection pressures in pregnant women. An investigation of relationships between rate of infection, injection pressures and extent of analgesia. Br J Anaesth. 1980 Jan;52(1):55-60. doi: 10.1093/bja/52.1.55. PMID 7378230
- [Background] Beilin Y, Bernstein HH, Zucker-Pinchoff B. The optimal distance that a multiorifice epidural catheter should be threaded into the epidural space. Anesth Analg. 1995 Aug;81(2):301-4. doi: 10.1097/00000539-199508000-00016. PMID 7618719
- [Result] de la Chapelle A, Carles M, Gleize V, Dellamonica J, Lallia A, Bongain A, Raucoules-Aime M. Impact of walking epidural analgesia on obstetric outcome of nulliparous women in spontaneous labour. Int J Obstet Anesth. 2006 Apr;15(2):104-8. doi: 10.1016/j.ijoa.2005.07.002. Epub 2006 Jan 24. PMID 16434183
- [Result] Apostolou GA, Zarmakoupis PK, Mastrokostopoulos GT. Spread of epidural anesthesia and the lateral position. Anesth Analg. 1981 Aug;60(8):584-6. PMID 7196172
- [Result] Grundy EM, Rao LN, Winnie AP. Epidural anesthesia and the lateral position. Anesth Analg. 1978 Jan-Feb;57(1):95-7. doi: 10.1213/00000539-197801000-00017. PMID 564647
- [Result] Beilin Y, Abramovitz SE, Zahn J, Enis S, Hossain S. Improved epidural analgesia in the parturient in the 30 degree tilt position. Can J Anaesth. 2000 Dec;47(12):1176-81. doi: 10.1007/BF03019865. PMID 11132738
- [Result] Shapiro A, Fredman B, Zohar E, Olsfanger D, Abu-Ras H, Jedeikin R. Alternating patient position following the induction of obstetric epidural analgesia does not affect local anaesthetic spread. Int J Obstet Anesth. 1998 Jul;7(3):153-6. doi: 10.1016/s0959-289x(98)80002-2. PMID 15321207